CLINICAL TRIAL: NCT05849740
Title: A Multicenter, Single-arm Exploratory Study of CD38 (Daratumumab) Monoclonal Antibody (Daratumumab) Combined Corticosteroid in the Treatment of Acquired Hemophilia A (AHA)
Brief Title: An Exploratory Study of Cluster of Differentiation 38 (CD38) Monoclonal Antibody Combined Corticosteroid in Acquired Hemophilia A
Acronym: AHA2023
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023013
Record Dates: First submitted 2023-04-18; First posted 2023-05-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Acquired Hemophilia
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Daratumumab and corticosteroid treatment
  Interventions: Drug: Daratumumab and corticosteroid treatment

INTERVENTIONS:
Drug: Daratumumab and corticosteroid treatment — Daratumumab and corticosteroid treatment
  Other Names: Intervention arm

SUMMARY:
To evaluate the time of response, sustained remission rate and relapse rate of CD38 monoclonal antibody (Daratumumab) combined corticosteroid in the treatment of AHA. To evaluate the safety of CD38 monoclonal antibody in the treatment of AHA.

DETAILED DESCRIPTION:
This is a prospective ,single-arm, multi-center controlled pilot trial of CD38 (Daratumumab) monoclonal antibody combined corticosteroid in the treatment of AHA patients.

Patients will receive Daratumumab and corticosteroid treatment in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all enrollment criteria before they can be enrolled:

Diagnosed as AHA; Women are postmenopausal women or women of childbearing age with strict contraception; Patients with good compliance

Exclusion Criteria:

* Patients with any of the following items cannot be enrolled in this study:

Congenital hemophilia with inhibitor; Pregnant and lactating women; Who are positive for hepatitis B surface antigen, hepatitis C antibody, HIV antibody (Ⅰ + Ⅱ) and syphilis antibody; Patients with poor compliance; Who cannot use contraception during the trial; Researchers believe that it is not appropriate for patients to participate in any other condition of this trial; Four weeks before entering the group, the patients received immunosuppressive therapy and the inhibitor showed a progressive decreasing trend (the change was less than 50%).

Acquired von Willebrand disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Total response rate to treatment (OR) Total response rate to treatment | During 8 weeks
  The proportion of patients achieving OR including CR and PR

SECONDARY OUTCOMES:
the proportion of patients with complete remission (CR) | During 8 weeks
  The proportion of patients achieving CR , which is defined as titer FVIII inhibitor lower than 0.6 Bethesda unit, factor VIII level≥ 50%
the proportion of patients with partial remission rate (PR) | During 8 weeks
  The proportion of patients achieving PR, which is defined as titer FVIII inhibitor higher than 0.6 Bethesda unit and factor VIII level≥ 50%, and no bleedings will be evaluated.
time to CR | During 8 weeks
  The time for patients to reach complete remission
The proportion of patients remaining in CR during 24 weeks | During 24 weeks
  The proportion of patients who reached CR and remain in CR during 24 weeks of follow -up time
The proportion of patients relapse after reaching CR during 24 weeks | During 24 weeks
  The proportion of patients who reached CR and relapse during 24 weeks of follow -up time
Safety outcome | From start of the treatment until the end of 24 weeks in the follow-up period
  Adverse events will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be requested from the corresponding authors from 12 months to 36 months after study completion
Supporting Information: Study Protocol
Time Frame: from 12 months to 36 months after study completion
Access Criteria: From corresponding author